CLINICAL TRIAL: NCT02016573
Title: Renal Denervation for Uncontrolled Hypertension
Acronym: RDNP-2012-02
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled into study and protocol has been superseded
Sponsor: Baker Heart and Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 070/12; 1034397 (Other Grant/Funding Number: NHMRC)
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Hypertension
Keywords: renal denervation; blood pressure; cardiovascular risk; target organ damage; sympathetic activity
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): participants randomised to the usual care group will receive additional antihypertensive medication in an attempt to achieve blood pressure targets
- Renal Denervation Group (Experimental): participants randomised to undergo the renal denervation procedure
  Interventions: Device: Renal Denervation

INTERVENTIONS:
Device: Renal Denervation — Renal Denervation Catheter
  Other Names: Symplicity Renal Denervation Catheter
  Arms: Renal Denervation Group

SUMMARY:
This is a study investigating the safety and usefulness of the Renal Denervation Procedure in reducing high blood pressure in people whose blood pressure is not adequately controlled despite already being treated with 2 blood pressure lowering drugs. This study is designed to compare the effects renal denervation to a usual care group.

DETAILED DESCRIPTION:
This is a phase 4 randomised control trial of renal denervation for the treatment of uncontrolled hypertension.

Previous studies have shown that the renal denervation procedure is safe and effective in reducing blood pressure.

A total of 100 participants with uncontrolled blood pressure, treated with two blood pressure lowering medications will be recruited into the study. Patients will be assigned to one of two groups. Participants in Group 1 will be assigned to undergo the renal denervation procedure. Participants in group 2 will undergo usual care, receiving additional antihypertensive medication in an attempt to reach blood pressure targets.

The duration of this study is 36 months.

ELIGIBILITY:
Inclusion Criteria:

* BP ≥140/90 mmHg (or ≥130/80 mmHg for patients with diabetes)
* concurrent treatment with 2 anti-hypertensive drugs

Exclusion Criteria:

* renal artery anatomy ineligible for treatment
* eGFR <15mL/min/1.73m2 (using MDRD formula)
* individual has had myocardial infarction, unstable angina or cerebrovascular accident within 6 months of screening visit
* female participants of child bearing potential must have negative pregnancy test prior to treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12 (Estimated); Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
blood pressure control | 6 months post procedure
  percentage of patients who achieve BP target at 6 months post intervention

SECONDARY OUTCOMES:
number of drugs required to reach target blood pressure | baseline to 6 months
  number of drugs required to reach target blood pressure
time to achieve blood pressure target | baseline to 6 months
  time to achieve blood pressure target
change in sympathetic nerve activity | baseline to 6 months
  changes in muscle sympathetic nerve activity (MSNA), renal and whole body Noradrenaline (NA) spillover
Change in left ventricular function | baseline to 6 months
  Change in left Ventricular ejection fraction, diastolic filling
Change in Quality of Life | baseline to 6 months
  Change in Quality of life as assessed be relevant questionnaires
Change in Serum Biochemistry | baseline to 6 months
  Plasma Renin Activity, aldosterone levels, estimated Glomerular Filtration Rate(eGFR), inflammatory markers, fasting glucose, fasting insulin, C-peptide, Homeostasis Model Assessment (HOMA) index, Lipid profile
Change in markers of arterial stiffness | baseline to 6 months
  Change in markers of arterial stiffness as assessed by Augmentation Index (AI) and Pulse Wave Velocity (PWV)
Change in left ventricular structure | baseline to 6 months
  Change in left ventricular mass index
Change in Urine Biochemistry | baseline to 6 months
  Urinary albumin creatinine ratio (UACR), 24 hour urinary creatinine clearance, sodium

CONTACTS AND LOCATIONS:
Overall Officials: Markus P Schlaich, MD, Principal Investigator — Baker IDI Heart & Diabetes Institute

IPD SHARING:
Plan to Share IPD: No
No data available